CLINICAL TRIAL: NCT03764995
Title: The Effects of Abdominal Massage on Functional (Primary) Chronic Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SERAP ÖZGÜL, Doc. Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-261/2018-32
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Constipation
Keywords: massage; abdominal massage; chronic constipation; primary constipation; functional constipation; defecation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal Massage (Experimental)
  Interventions: Other: Standard bowel management; Other: Abdominal massage
- Placebo Ultrasound (Placebo Comparator)
  Interventions: Other: Standard bowel management; Other: Placebo Ultrasound

INTERVENTIONS:
Other: Standard bowel management — Lifestyle advices such as increasing fluid and fibre intake, improving physical activity level, and taking the ideal posture for defecation (squatting position) with a two-pages document.
Other: Abdominal massage — Abdominal massage will be performed three days a week for four weeks. Each session will last around 15-20 minutes.
  Arms: Abdominal Massage
Other: Placebo Ultrasound — Placebo ultrasound (US) will be applied to the abdominal region for four weeks, 2 days of the week and 15 minutes per day.
  Arms: Placebo Ultrasound

SUMMARY:
The aim of the present study is to investigate the efficacy of abdominal massage in patients with functional (primary) chronic constipation. The present study is designed as a randomized placebo controlled. Since the placebo group is included in the research design, if there is a greater improvement of symptoms of constipation and quality of life in the massage group when compared to the control group, it will be determined that this effect is not related to a placebo effect. If the efficacy of Abdominal Massage is revealed with a placebo controlled design, the therapist effect will be eliminated and further evidence on a well-known massage technique in functional (primary) chronic constipation, a common gastrointestinal problem, will be provided. The results of the present placebo controlled randomized trial will indicate that the need for pharmacological agents and the side effects associated with these agents will be reduced. According to the literature, there are studies that investigate the effects of abdominal massage on symptoms of constipation and quality of life. However, it has generally been used for secondary constipation or two applications have been compared. In addition, there is no randomized placebo-controlled study investigating the effect of abdominal massage on severity of chronic constipation and quality of life.

DETAILED DESCRIPTION:
Constipation is a subjective symptom that defines as inadequate defecation including several symptoms as follows: the sensation of incomplete bowel evacuation, hard stool, straining, and difficulty in defecation. The general prevalence of constipation in adults is 16%. The pre-defined risk factors are women gender, advanced age, non-white ethnicity, low socio-economic level, decreased physical activity underlying diseases, and medications. Chronic constipation affects quality of life and causes problems such as anxiety, depression, somatization, sleep disorders, sexual dysfunctions, school/work absenteeism. In the following periods, it causes serious comorbidities including dyspnea, gastro-esophageal reflux, hypertension, thyroid diseases, vaginitis, dyspareunia, diabetes, and fibromyalgia.

In the treatment of chronic constipation, conservative approaches (lifestyle change and physiotherapy applications) are used at the first phase. If conservative approaches are not helpful for patients pharmacological and surgical treatment can be performed based on the characteristics of patients, respectively. Pharmacological treatments aim to increase the frequency of spontaneous bowel movements, to reduce abdominal pain and swelling, and to improve stool consistency. However, side effects such as abdominal bloating, abdominal cramping, abdominal pain, stomach gas, nausea, diarrhea, headache and dyspnea are reported by patients in the following period. Furthermore, medications for constipation management are not cost-effective. Therefore, the level of evidence on conservative approaches with low cost, non-invasive and no-side effects in constipation treatment should be increased.

Physiotherapy approaches to alleviate chronic constipation symptoms include such as defecation training, abdominal massage, connective tissue massage, electrical stimulation, Kinesio-taping, anorectal biofeedback, and exercise training. Abdominal massage application in constipation is used in constipation management since the early 1870s and it is popular in recent years. The benefits of abdominal massage are known as follows: reduction in the abdominal muscle tension, improvement of local circulation, and stimulation of peristaltic movements. The technique of abdominal massage consists of 5 stages as follows: abdominal muscle stroking, colon stroking, colon kneading, colon stroking, and abdominal muscle stroking.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Diagnosed with chronic constipation according to Rome IV criteria

Exclusion Criteria:

* A recent history of abdominal surgery
* Intestinal obstruction, ileus, colon cancer
* Enteric neuropathic patients: Diabetic intestinal neuropathy, Hirschsprung's disease, Megacolon, Megarectum
* Umbilical hernia
* Metabolic diseases: Cancer, Chronic renal failure, Severe cardiovascular disease, Hepatic failure, Hepatosplenomegaly, Abdominal aortic aneurysm
* Neurological diseases: Parkinson, Spinal cord injury, Multiple sclerosis, Cerebro-vascular event,
* Paraplegia Mental problem to prevent co-operative treatment
* Pregnancy and lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Severity of constipation | Change in severity of constipation from baseline at 4 weeks
  Constipation Severity Instrument (CSI) will be used to evaluate the severity of the constipation. CSI was designed to evaluate defecation frequency and consistency as well as the level of straining experienced by individuals during bowel movement. There are three subscales of CSI, obstructive defecation (OT), colonic inertia (CI), and pain. Higher scores of CSI indicate more severe constipation.

SECONDARY OUTCOMES:
Patient Assessment of Constipation Quality of life | Change in quality of life from baseline at 4 weeks
  Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QOL) will be used to evaluate quality of life. This questionnaire includes a total of 28 items in 4 subscales: worries and concerns (11 items), physical discomfort (4 items), psychosocial discomfort (8 items), and satisfaction (5 items). Higher scores of PAC-QOL indicate more negative effects of constipation on the quality of life.
Stool consistency | Change from baseline stool consistency at 4 weeks
  The stool consistency will be evaluated using the Bristol Stool Scale (BSS), quick and useful indicator of the colonic transit time , a seven-point scale (from 1 to 7), type 1=separate hard lumps, like nuts; 2=sausage shaped but lumpy; 3=like a sausage or snake, but with cracks on its surface; 4=like a sausage or snake, smooth and soft; 5=soft blobs with clear cut edges; 6=pieces with ragged edges, a mushy stool; 7=water, no solid pieces. While type 1 and 2 indicate hard stool, type 3,4 and 5 show looser (ideal) stool.
Symptoms of constipation | Change from baseline symptoms of constipation at 4 weeks
  In order to gather information regarding the participants' symptoms of constipation, they will be asked to complete a 7-day bowel diary during the treatment period. This diary includes items regarding the frequency of bowel movement, stool consistency, defecation time, feeling of incomplete evacuation, and changes in food and liquid consumption.
Abdominal pain, abdominal bloating severity and the effect of life | Change from baseline symptoms of constipation at 4 weeks
  Visual Analogue Scale (VAS): This scale is a 10 cm horizontal line. 0 = no pain / bloating / meaning no effect, 10 = unbearable pain / bloating / experiencing
Physical activity levels | Change from baseline symptoms of constipation at 4 weeks
  The physical activity levels of the individuals in the last seven days are evaluated under 4 headings (severe activities, moderate activity, walking and sitting). While calculating the total score, the MET-min scores of the patients are obtained by multiplying the duration of activity and frequency of activities (number of days) by the BAT values given to activities (severe activity = 8 MET, moderate activity = 4 MET, walking = 3.3 MET)
Patient global change scale | Change from baseline patient global change at 4 weeks
  It is a 7-item scale that evaluates the perception of the change in the effect of constipation and related complaints on the life of the patient compared to the study. The options on this scale are ''much much better'', ''much better'', 'a little better'', ''no change", ''a little worse'', ''much worse'', ''much much worse''

CONTACTS AND LOCATIONS:
Locations (1):
- Ceren Gursen, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lamas K, Lindholm L, Stenlund H, Engstrom B, Jacobsson C. Effects of abdominal massage in management of constipation--a randomized controlled trial. Int J Nurs Stud. 2009 Jun;46(6):759-67. doi: 10.1016/j.ijnurstu.2009.01.007. Epub 2009 Feb 12. PMID 19217105
- [Background] Sinclair M. The use of abdominal massage to treat chronic constipation. J Bodyw Mov Ther. 2011 Oct;15(4):436-45. doi: 10.1016/j.jbmt.2010.07.007. Epub 2010 Aug 25. PMID 21943617
- [Background] Lamas K, Graneheim UH, Jacobsson C. Experiences of abdominal massage for constipation. J Clin Nurs. 2012 Mar;21(5-6):757-65. doi: 10.1111/j.1365-2702.2011.03946.x. Epub 2011 Nov 21. PMID 22098585
- [Derived] Dogan IG, Gursen C, Akbayrak T, Balaban YH, Vahabov C, Uzelpasaci E, Ozgul S. Abdominal Massage in Functional Chronic Constipation: A Randomized Placebo-Controlled Trial. Phys Ther. 2022 Jul 4;102(7):pzac058. doi: 10.1093/ptj/pzac058. PMID 35554601